CLINICAL TRIAL: NCT01318135
Title: A Long-term, Open-label Extension Study to Investigate the Long-term Safety of Alogliptin When Used in Combination With Sulfonylurea or Metformin in Subjects With Type 2 Diabetes in Japan
Brief Title: Long-term Safety Study of Alogliptin Used in Combination With Sulfonylurea or Metformin in Participants With Type 2 Diabetes in Japan
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYR-322/OCT-005; JapicCTI-090902 (Registry Identifier: JapicCTI); U1111-1119-6196 (Registry Identifier: WHO)
Record Dates: First submitted 2011-03-16; First posted 2011-03-18 (Estimated); Results first posted 2012-08-16 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus - Type 2; Diabetes Mellitus; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — alogliptin; glimepiride; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID (Active Comparator)
  Interventions: Drug: Alogliptin and glimepiride
- Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID (Active Comparator)
  Interventions: Drug: Alogliptin and glimepiride
- Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID (Active Comparator)
  Interventions: Drug: Alogliptin and metformin
- Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID (Active Comparator)
  Interventions: Drug: Alogliptin and metformin

INTERVENTIONS:
Drug: Alogliptin and glimepiride — Alogliptin 12.5 mg, tablets, orally, once daily and sulfonylurea 1, 2, 3, 4, 5 or 6 mg, tablets, orally, once or twice daily for up to 52 weeks.
  Other Names: SYR-322; Amaryl
  Arms: Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID
Drug: Alogliptin and glimepiride — Alogliptin 25 mg, tablets, orally, once daily and sulfonylurea 1, 2, 3, 4, 5 or 6 mg, tablets, orally, once or twice daily for up to 52 weeks.
  Other Names: SYR-322; Amaryl
  Arms: Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID
Drug: Alogliptin and metformin — Alogliptin 12.5 mg, tablets, orally, once daily and metformin 500 mg, tablets, orally, twice daily or metformin 750 mg, tablets, orally, three times daily for up to 52 weeks.
  Other Names: SYR-322; Glycoran
  Arms: Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID
Drug: Alogliptin and metformin — Alogliptin 25 mg, tablets, orally, once daily and metformin 500 mg, tablets, orally, twice daily or metformin 750 mg, tablets, orally, three times daily for up to 52 weeks.
  Other Names: SYR-322; Glycoran
  Arms: Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID

SUMMARY:
To evaluate the efficacy and safety of alogliptin administered as an add-on to sulfonylurea (glimepiride) or metformin, once daily (QD), twice daily (BID) or three times daily (TID).

DETAILED DESCRIPTION:
Both insulin hyposecretion and insulin-resistance are considered to be involved in the development of type 2 diabetes mellitus.

Takeda is developing SYR-322 (alogliptin) for the improvement of glycemic control in patients with type 2 diabetes mellitus. Alogliptin is an inhibitor of the dipeptidyl peptidase IV (DPP-IV) enzyme. DPP-IV is thought to be primarily responsible for the degradation of 2 peptide hormones released in response to nutrient ingestion. It is expected that inhibition of DPP-IV will improve glycemic control in patients with type 2 diabetes.

This was a phase 2/3, multicenter, open-label study, in participants who had completed the core phase 2/3 sulfonylurea add-on study (SYR-322/CCT-005; NCT01318083) or the core phase 2/3 metformin add-on study (SYR-322/CCT-006; NCT01318109) to evaluate the safety and efficacy of alogliptin administered as an add-on to a sulfonylurea (glimepiride) or metformin continuously for 40 weeks (52 weeks from the start of study treatment with alogliptin in the core phase 2/3 sulfonylurea add-on study or the core phase 2/3 metformin add-on study).

ELIGIBILITY:
Inclusion Criteria:

Common criteria that applied to participants completing both the core phase 2/3 sulfonylurea add-on study and those completing the core phase 2/3 metformin add-on study:

1. Had completed the core phase 2/3 sulfonylurea add-on study or the core phase 2/3 metformin add-on study.
2. Was capable of understanding and complying with protocol requirements.
3. Signed a written informed consent form prior to the initiation of any study procedure.

Exclusion Criteria:

Common criteria that applied to participants completing both the core phase 2/3 sulfonylurea add-on study and those completing the core phase 2/3 metformin add-on study:

1. With clinical manifestation of hepatic impairment (eg, an aspartate aminotransferase or alanine aminotransferase value of 2.5 times or more of the upper reference limit at Week 8 of the core phase 2/3 sulfonylurea add-on study or the core phase 2/3 metformin add-on study).
2. With clinical manifestation of renal impairment (eg, a creatinine value of 1.5 times or more of the upper reference limit at Week 8 of the core phase 2/3 sulfonylurea add-on study or the core phase 2/3 metformin add-on study).
3. With serious cardiac disease, cerebrovascular disorder, or serious pancreatic or hematological disease (eg, a subject who requires hospital admission).

Criteria that applied only to participants completing the core phase 2/3 metformin add-on study:

1. With history or symptoms of lactic acidosis.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 576 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Diabetes and Endocrine Division, Study Director — Department of Medicine, Kawasaki Medical School

REFERENCES:
- [Derived] Seino Y, Hiroi S, Hirayama M, Kaku K. Efficacy and safety of alogliptin added to sulfonylurea in Japanese patients with type 2 diabetes: A randomized, double-blind, placebo-controlled trial with an open-label, long-term extension study. J Diabetes Investig. 2012 Dec 20;3(6):517-25. doi: 10.1111/j.2040-1124.2012.00226.x. Epub 2012 Jul 12. PMID 24843617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 58 investigative sites in Japan from 06 January 2009 to 23 January 2010.
Pre-assignment Details: Participants who had completed a core phase 2/3 glimepiride (SYR-322/CCT-005; NCT01318083) or metformin (SYR-322/CCT-006; NCT01318109) add-on study were enrolled in one of four, once daily (QD) or twice-daily (BID) treatment groups. Five participants completed OCT-005 study without receiving the study drug.
Groups:
- CCT/005 - 12.5 mg Dose Group* → 12.5 mg Combination Group: Alogliptin 12.5 mg, tablets, orally, once daily and glimepiride 1, 2, 3, 4, 5 or 6 mg, tablets, orally, once or twice daily for up to 52 weeks.
  *for participants from the 12.5 mg combination dosing ARM of the SYR-322/CCT-005 (NCT01318083) core phase 2/3 glimepiride add-on study.
- CCT/005 - 25 mg Dose Group* → 25 mg Combination Dose Group: Alogliptin 25 mg, tablets, orally, once daily and glimepiride 1, 2, 3, 4, 5 or 6 mg, tablets, orally, once or twice daily for up to 52 weeks.
  *for participants from the 25 mg combination dosing ARM of the SYR-322/CCT-005 (NCT01318083) core phase 2/3 glimepiride add-on study.
- Glimepiride Monotherapy Group* → 12.5 mg Combination Group: Alogliptin 12.5 mg, tablets, orally, once daily and glimepiride 1, 2, 3, 4, 5 or 6 mg, tablets, orally, once or twice daily for up to 52 weeks.
  *for participants from the glimepiride 1, 2, 3 or 4 mg dosing ARM of the SYR-322/CCT-005 (NCT01318083) core phase 2/3 glimepiride add-on study.
- Glimepiride Monotherapy Group* → 25 mg Combination Group: Alogliptin 25 mg, tablets, orally, once daily and glimepiride 1, 2, 3, 4, 5 or 6 mg, tablets, orally, once or twice daily for up to 52 weeks.
  *for participants from the glimepiride 1, 2, 3 or 4 mg dosing ARM of the SYR-322/CCT-005 (NCT01318083) core phase 2/3 glimepiride add-on study.
- CCT/006 - 12.5 mg Dose Group* → 12.5 mg Combination Group: Alogliptin 12.5 mg, tablets, orally, once daily and metformin 500 mg, tablets, orally, twice daily or metformin 750 mg, tablets, orally, three times daily for up to 52 weeks.
  *for participants from the 12.5 mg combination dosing ARM of the SYR-322/CCT-006 (NCT01318109) core phase 2/3 metformin add-on study.
- CCT/006 - 25 mg Dose Group* → 25 mg Combination Group: Alogliptin 25 mg, tablets, orally, once daily and metformin 500 mg, tablets, orally, twice daily or metformin 750 mg, tablets, orally, three times daily for up to 52 weeks.
  *for participants from the 25 mg combination dosing ARM of the SYR-322/CCT-006 (NCT01318109) core phase 2/3 metformin add-on study.
- Metformin Monotherapy Group* → 12.5 mg Combination Group: Alogliptin 12.5 mg, tablets, orally, once daily and metformin 500 mg, tablets, orally, twice daily or metformin 750 mg, tablets, orally, three times daily for up to 52 weeks.
  *for participants from the metformin 500 mg or 750 mg dosing ARM of the SYR-322/CCT-006 (NCT01318109) core phase 2/3 metformin add-on study.
- Metformin Monotherapy Group* → 25 mg Combination Group: Alogliptin 25 mg, tablets, orally, once daily and metformin 500 mg, tablets, orally, twice daily or metformin 750 mg, tablets, orally, three times daily for up to 52 weeks.
  *for participants from the metformin 500 mg or 750 mg dosing ARM of the SYR-322/CCT-006 (NCT01318109) core phase 2/3 metformin add-on study.
Period: Enrolled - Long-Term Extension Study
Arm/Group | CCT/005 - 12.5 mg Dose Group* → 12.5 mg Combination Group | CCT/005 - 25 mg Dose Group* → 25 mg Combination Dose Group | Glimepiride Monotherapy Group* → 12.5 mg Combination Group | Glimepiride Monotherapy Group* → 25 mg Combination Group | CCT/006 - 12.5 mg Dose Group* → 12.5 mg Combination Group | CCT/006 - 25 mg Dose Group* → 25 mg Combination Group | Metformin Monotherapy Group* → 12.5 mg Combination Group | Metformin Monotherapy Group* → 25 mg Combination Group
Started | 99 | 102 | 46 | 49 | 91 | 90 | 50 | 49
Completed | 97 | 102 | 46 | 49 | 91 | 90 | 50 | 49
Not Completed | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Treatment Complications | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Entered - Long-Term Extension Study
Arm/Group | CCT/005 - 12.5 mg Dose Group* → 12.5 mg Combination Group | CCT/005 - 25 mg Dose Group* → 25 mg Combination Dose Group | Glimepiride Monotherapy Group* → 12.5 mg Combination Group | Glimepiride Monotherapy Group* → 25 mg Combination Group | CCT/006 - 12.5 mg Dose Group* → 12.5 mg Combination Group | CCT/006 - 25 mg Dose Group* → 25 mg Combination Group | Metformin Monotherapy Group* → 12.5 mg Combination Group | Metformin Monotherapy Group* → 25 mg Combination Group
Started | 97 (Patients participated in CCT-005 but not entered OCT-005 are excluded in Participant Flow.) | 102 (Patients participated in CCT-005 but not entered OCT-005 are excluded in Participant Flow.) | 46 (Patients participated in CCT-005 but not entered OCT-005 are excluded in Participant Flow.) | 49 (Patients participated in CCT-005 but not entered OCT-005 are excluded in Participant Flow.) | 90 (Patients participated in CCT-006 but not entered OCT-005 are excluded in Participant Flow.) | 87 (Patients participated in CCT-006 but not entered OCT-005 are excluded in Participant Flow.) | 50 (Patients participated in CCT-006 but not entered OCT-005 are excluded in Participant Flow.) | 49 (Patients participated in CCT-006 but not entered OCT-005 are excluded in Participant Flow.)
Completed | 80 (296 participants enrolled and 294 completed glimepiride add-on study and entered the present study.) | 89 (296 participants enrolled and 294 completed glimepiride add-on study and entered the present study.) | 38 (296 participants enrolled and 294 completed glimepiride add-on study and entered the present study.) | 42 (296 participants enrolled and 294 completed glimepiride add-on study and entered the present study.) | 81 (280 participants enrolled and 276 completed metformin add-on study and entered the present study.) | 83 (280 participants enrolled and 276 completed metformin add-on study and entered the present study.) | 49 (280 participants enrolled and 276 completed metformin add-on study and entered the present study.) | 46 (280 participants enrolled and 276 completed metformin add-on study and entered the present study.)
Not Completed | 17 | 13 | 8 | 7 | 9 | 4 | 1 | 3
Not completed — Adverse Event | 9 | 3 | 4 | 3 | 4 | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 2 | 1 | 2 | 0 | 0 | 1
Not completed — Lack of Efficacy | 5 | 7 | 2 | 3 | 2 | 2 | 1 | 1
Not completed — Use of Excluded Medications | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID: Alogliptin 12.5 mg, tablets, orally, once daily and sulfonylurea 1, 2, 3, 4, 5 or 6 mg, tablets, orally, once or twice daily for up to 52 weeks.
- Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID: Alogliptin 25 mg, tablets, orally, once daily and sulfonylurea 1, 2, 3, 4, 5 or 6 mg, tablets, orally, once or twice daily for up to 52 weeks.
- Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID: Alogliptin 12.5 mg, tablets, orally, once daily and metformin 500 mg, tablets, orally, twice daily or metformin 750 mg, tablets, orally, three times daily for up to 52 weeks.
- Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID: Alogliptin 25 mg, tablets, orally, once daily and metformin 500 mg, tablets, orally, twice daily or metformin 750 mg, tablets, orally, three times daily for up to 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID | Total
Number analyzed (Participants) | 150 | 152 | 142 | 145 | 589
Age, Customized [Number; unit: participants] — Participants randomized in core phase 2/3 glimepiride add-on study, excluding those randomized to the "glimepiride monotherapy group" was 304. Participants randomized in core phase 2/3 metformin add-on study, excluding those randomized to the "metformin monotherapy group" was 287. The following are included in baseline: Column 1: 7 patients participated in CCT-005 but not entered OCT-005; Column 2: 1 participated in CCT-005 but not entered OCT-005; Column 3: 2 participated in CCT-006 but not entered OCT-005; Column 4: 9 participated in CCT-006 but not entered OCT-005.
  participants
    ≤ 64 years | 93 (9.50) | 105 (8.92) | 142 (8.12) | 145 (8.41) | 485
    ≥ 65 years | 57 | 47 | 0 | 0 | 104
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 52 | 46 | 44 | 195
  Male | 97 | 100 | 96 | 101 | 394

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events.
Description: Treatment-emergent adverse events (TEAE) are defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through 30 days after receiving the last dose of study drug. A TEAE may also be a pretreatment adverse event or a concurrent medical condition diagnosed prior to the date of first dose of study drug that increases in severity after the start of dosing.
Time Frame: 52 Weeks.
Population: Full Analysis Set was defined as the population of participants randomized in the core phase 2/3 SYR-322/CCT-005 (NCT01318083) or SYR-322/CCT-006 (NCT01318109) add-on studies and received at least 1 dose of the investigational products (SYR-322DB in combination with glimepiride or metformin) for the treatment period were identified for analysis.
Measure: Number; unit: participants
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 150 | 152 | 142 | 145
participants
  Serious Adverse Event | 16 | 3 | 7 | 5
  Other Adverse Event (≥3% Frequency Threshold) | 116 | 134 | 108 | 113

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 8).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 8 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 8.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 147 | 150 | 141 | 143
percentage of Glycosylated Hemoglobin | -0.53 (0.506) | -0.65 (0.515) | -0.53 (0.486) | -0.59 (0.394)

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 12).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 12 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 145 | 148 | 140 | 142
percentage of Glycosylated Hemoglobin | -0.63 (0.626) | -0.72 (0.589) | -0.61 (0.576) | -0.71 (0.489)

4. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 16).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 16 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 16.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 141 | 147 | 138 | 135
percentage of Glycosylated Hemoglobin | -0.66 (0.685) | -0.76 (0.660) | -0.69 (0.614) | -0.78 (0.495)

5. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 20).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 20 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 20.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 139 | 146 | 136 | 134
percentage of Glycosylated Hemoglobin | -0.63 (0.754) | -0.70 (0.689) | -0.67 (0.648) | -0.78 (0.553)

6. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 24).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 24 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 24.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 137 | 145 | 135 | 134
percentage of Glycosylated Hemoglobin | -0.59 (0.823) | -0.70 (0.740) | -0.68 (0.668) | -0.78 (0.623)

7. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 28).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 28 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 28.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 132 | 144 | 135 | 132
percentage of Glycosylated Hemoglobin | -0.62 (0.841) | -0.76 (0.721) | -0.70 (0.659) | -0.84 (0.596)

8. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 32).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 32 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 32.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 132 | 140 | 135 | 129
percentage of Glycosylated Hemoglobin | -0.63 (0.868) | -0.77 (0.736) | -0.67 (0.644) | -0.81 (0.634)

9. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 36).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 36 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 36.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 128 | 137 | 134 | 129
percentage of Glycosylated Hemoglobin | -0.64 (0.881) | -0.77 (0.745) | -0.67 (0.659) | -0.79 (0.653)

10. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 40).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 40 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 40.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 124 | 135 | 132 | 129
percentage of Glycosylated Hemoglobin | -0.66 (0.799) | -0.74 (0.779) | -0.63 (0.676) | -0.74 (0.698)

11. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 44).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 44 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 44.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 84 | 90 | 81 | 83
percentage of Glycosylated Hemoglobin | -0.48 (0.726) | -0.71 (0.666) | -0.47 (0.787) | -0.70 (0.688)

12. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 48).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 48 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 48.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 82 | 90 | 81 | 83
percentage of Glycosylated Hemoglobin | -0.40 (0.706) | -0.61 (0.660) | -0.36 (0.762) | -0.62 (0.707)

13. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 52).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 52 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 52.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 80 | 89 | 81 | 83
percentage of Glycosylated Hemoglobin | -0.33 (0.652) | -0.53 (0.643) | -0.29 (0.744) | -0.53 (0.790)

14. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Final Visit).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at final visit and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Final Visit (up to 52).
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 149 | 152 | 142 | 145
percentage of Glycosylated Hemoglobin | -0.42 (0.838) | -0.58 (0.791) | -0.44 (0.720) | -0.58 (0.781)

15. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 8).
Description: The change between the value of fasting blood glucose collected at week 8 and baseline.
Time Frame: Baseline and Week 8.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 147 | 150 | 141 | 143
mg/dL | -20.7 (26.50) | -19.6 (30.53) | -22.0 (22.76) | -23.4 (26.75)

16. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 12).
Description: The change between the value of fasting blood glucose collected at week 12 and baseline.
Time Frame: Baseline and Week 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 145 | 148 | 140 | 142
mg/dL | -22.0 (32.19) | -18.1 (29.05) | -22.9 (24.04) | -24.2 (27.30)

17. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 16).
Description: The change between the value of fasting blood glucose collected at week 6 and baseline.
Time Frame: Baseline and Week 16.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 141 | 147 | 138 | 135
mg/dL | -22.3 (34.37) | -17.8 (32.22) | -21.8 (26.86) | -26.1 (26.93)

18. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 20).
Description: The change between the value of fasting blood glucose collected at week 20 and baseline.
Time Frame: Baseline and Week 20.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 139 | 146 | 136 | 134
mg/dL | -22.4 (31.75) | -22.3 (30.93) | -23.4 (27.88) | -26.1 (26.19)

19. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 24).
Description: The change between the value of fasting blood glucose collected at week 24 and baseline.
Time Frame: Baseline and Week 24.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 137 | 145 | 135 | 133
mg/dL | -24.0 (31.69) | -25.0 (32.68) | -25.6 (24.22) | -26.3 (28.09)

20. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 28).
Description: The change between the value of fasting blood glucose collected at week 28 and baseline.
Time Frame: Baseline and Week 28.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 132 | 144 | 135 | 131
mg/dL | -19.9 (36.87) | -25.9 (33.67) | -25.8 (26.16) | -28.2 (29.49)

21. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 32).
Description: The change between the value of fasting blood glucose collected at week 32 and baseline.
Time Frame: Baseline and Week 32.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 132 | 139 | 135 | 129
mg/dL | -22.4 (37.47) | -26.1 (30.69) | -23.2 (25.71) | -28.2 (29.31)

22. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 36).
Description: The change between the value of fasting blood glucose collected at week 36 and baseline.
Time Frame: Baseline and Week 36.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 128 | 136 | 134 | 129
mg/dL | -25.5 (34.16) | -26.7 (33.12) | -23.4 (24.00) | -26.0 (31.26)

23. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 40).
Description: The change between the value of fasting blood glucose collected at week 40 and baseline.
Time Frame: Baseline and Week 40.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 124 | 135 | 132 | 129
mg/dL | -21.3 (33.44) | -22.7 (30.19) | -19.8 (24.81) | -23.2 (31.13)

24. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 44).
Description: The change between the value of fasting blood glucose collected at week 44 and baseline.
Time Frame: Baseline and Week 44.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 83 | 90 | 81 | 83
mg/dL | -15.4 (31.69) | -21.9 (29.33) | -16.3 (26.22) | -24.0 (31.49)

25. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 48).
Description: The change between the value of fasting blood glucose collected at week 48 and baseline.
Time Frame: Baseline and Week 48.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 82 | 90 | 81 | 83
mg/dL | -13.6 (28.29) | -16.6 (30.68) | -14.3 (24.22) | -23.3 (29.73)

26. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Week 52).
Description: The change between the value of fasting blood glucose collected at week 52 and baseline.
Time Frame: Baseline and Week 52.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 80 | 89 | 81 | 83
mg/dL | -13.3 (31.74) | -11.9 (30.11) | -14.0 (26.92) | -16.1 (29.60)

27. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (Final Visit).
Description: The change between the value of fasting blood glucose collected at final visit and baseline.
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 149 | 152 | 141 | 145
mg/dL | -16.0 (33.73) | -13.0 (34.68) | -16.4 (25.81) | -17.7 (29.54)

28. Secondary Outcome: Change From Baseline in Blood Glucose Measured by the Meal Tolerance Test (Week 12).
Description: The change between the value of blood glucose measured by the meal tolerance test collected at week 12 and blood glucose measured by the meal tolerance test collected at baseline. Meal tolerance test measures blood glucose through blood samples drawn before a meal and at 2 hours after the start of the meal.
Time Frame: Baseline and Week 12.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 146 | 149 | 141 | 143
mg/dL | 80.2 (43.24) | 80.1 (47.77) | 61.6 (38.72) | 64.0 (34.39)

29. Secondary Outcome: Change From Baseline in Blood Glucose Measured by the Meal Tolerance Test (Week 24).
Description: The change between the value of blood glucose measured by the meal tolerance test collected at week 24 and blood glucose measured by the meal tolerance test collected at baseline. Meal tolerance test measures blood glucose through blood samples drawn before a meal and at 2 hours after the start of the meal.
Time Frame: Baseline and Week 24.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 97 | 101 | 85 | 84
mg/dL | 87.4 (38.74) | 77.9 (42.68) | 60.7 (34.96) | 62.4 (32.23)

30. Secondary Outcome: Change From Baseline in Blood Glucose Measured by the Meal Tolerance Test (Week 52).
Description: The change between the value of blood glucose measured by the meal tolerance test collected at week 52 and blood glucose measured by the meal tolerance test collected at baseline. Meal tolerance test measures blood glucose through blood samples drawn before a meal and at 2 hours after the start of the meal.
Time Frame: Baseline and Week 52.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 120 | 135 | 130 | 129
mg/dL | 83.8 (46.24) | 83.2 (43.61) | 62.5 (42.91) | 62.7 (32.81)

31. Secondary Outcome: Change From Baseline in Blood Glucose Measured by the Meal Tolerance Test (Final Visit).
Description: The change between the value of blood glucose measured by the meal tolerance test collected at final visit and blood glucose measured by the meal tolerance test collected at baseline. Meal tolerance test measures blood glucose through blood samples drawn before a meal and at 2 hours after the start of the meal.
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Number analyzed (Participants) | 146 | 149 | 141 | 143
mg/dL | 84.8 (45.47) | 84.9 (44.35) | 63.5 (43.06) | 63.7 (32.32)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through 30 days after receiving the last dose of study drug.
Description: The following are included in Adverse Events tables: Column 1: 7 patients participated in CCT-005 but not entered OCT-005; Column 2: 1 participated in CCT-005 but not entered OCT-005; Column 3: 2 participated in CCT-006 but not entered OCT-005; Column 4: 9 participated in CCT-006 but not entered OCT-005.
Arm/Group | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID
Serious Adverse Events (participants affected / at risk) | 16/150 | 3/152 | 7/142 | 5/145
Other Adverse Events (participants affected / at risk) | 116/150 | 134/152 | 108/142 | 113/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID (N=150) | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID (N=152) | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID (N=142) | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID (N=145)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0/0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Cerebral circulatory failure (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Embolic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Gas gangrene (Infections and infestations) | 1 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0/0 | 0 | 1
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0/1 | 1 | 0
Pneumonia legionella (Infections and infestations) | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 12.5 mg QD and Glimepiride 1- 6 mg QD or BID (N=150) | Alogliptin 25 mg QD and Glimepiride 1 - 6 mg QD or BID (N=152) | Alogliptin 12.5 mg QD and Metformin 500 mg BID or 750 mg TID (N=142) | Alogliptin 25 mg QD and Metformin 500 mg BID or 750 mg TID (N=145)
Alanine aminotransferase increased (Investigations) | 0 | 0 | 6 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 4 | 2 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 11 | 9 | 6
Blood creatine phosphokinase increased (Investigations) | 2 | 5 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 6
Cataract (Eye disorders) | 6 | 7 | 0 | 0
Chest pain (General disorders) | 1 | 5 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1 | 6
Constipation (Gastrointestinal disorders) | 7 | 7 | 7 | 8
Cystitis (Infections and infestations) | 5 | 5 | 5 | 4
Dental caries (Gastrointestinal disorders) | 6 | 1 | 1 | 7
Diabetic retinopathy (Eye disorders) | 4 | 8 | 6 | 10
Diarrhoea (Gastrointestinal disorders) | 5 | 3 | 6 | 3
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 7 | 6
Fall (Injury, poisoning and procedural complications) | 7 | 12 | 0 | 0
Gastritis (Gastrointestinal disorders) | 4 | 8 | 0 | 0
Gastroenteritis (Infections and infestations) | 7 | 4 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 9 | 3
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 2 | 5
Hypertension (Vascular disorders) | 0 | 0 | 7 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 8 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 5
Nasopharyngitis (Infections and infestations) | 46 | 57 | 44 | 53
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 1 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 7 | 4 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 10 | 16 | 6 | 6
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 5 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinical trial contract states that information should never be disclosed without prior consent of the sponsor, although it does not specify the number of days during which disclosure of information is limited.